CLINICAL TRIAL: NCT02830828
Title: How Does Disease Severity, Object Weight, Object Friction, and Sudden Changes to Object Weight Affect Precision Pinch Grip Force in Carpal Tunnel Syndrome?
Brief Title: Studying Finger-thumb Grip in Patients With Carpal Tunnel Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Thomas Edward Pidgeon (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor-Investigator, Thomas Edward Pidgeon, Chief Investigator, University Hospital Birmingham NHS Foundation Trust
Organization: University Hospital Birmingham NHS Foundation Trust (Other)
Other Study IDs: RRK5257
Record Dates: First submitted 2015-03-27; First posted 2016-07-13 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Patients fulfilling inclusion/exclusion criteria referred to the PI with suspected carpal tunnel syndrome.
  Interventions: Other: Investigation of precision pinch grip control
- Controls: Healthy volunteers fulfilling inclusion/exclusion criteria with no symptoms of carpal tunnel syndrome.
  Mid-study, it was elected to also match patients to their own contralateral disease-free hand to act as a control.
  Interventions: Other: Investigation of precision pinch grip control

INTERVENTIONS:
Other: Investigation of precision pinch grip control

SUMMARY:
INTRODUCTION Carpal tunnel syndrome (CTS) is a common condition that results in impaired hand function. In cases of CTS the "pinch grip" force between the thumb and index finger becomes unnecessarily high to prevent objects from slipping when they are picked up.

HYPOTHESES The proposed study will investigate the following hypotheses regarding CTS.

As an object is picked up, the investigators suspect there will be several points at which grip force will be different between patients with different severities of CTS, i.e. grip may deteriorate as CTS gets worse.

The investigators also suspect grip force will be affected depending on the weight of the object, i.e. patients with CTS may struggle with objects of a certain weight.

Patients with CTS sweat less, and this may affect their grip. The investigators suspect that pinch grip in CTS patients is disproportionately altered by the frictional properties of the object and by the moistness of the skin.

The investigators suspect patients with CTS will be less able to adapt to sudden changes in an object's weight.

The investigators wish to examine how the above are affected after surgical treatment of CTS.

METHODS The investigators will include patients with symptomatic, idiopathic CTS, aged between 18 and 80 years. The investigators' centre will recruit CTS patients who will attend their National Health Service (NHS) outpatient appointment followed by nerve conduction studies. An equal number of healthy participants will be recruited for comparison purposes.

At the aforementioned appointment, patients will undertake a pinch grip force test using a device that will test the above points.

Patients will have normal care under their surgeon, which may include an operation for treatment of CTS. Therefore some patients will be invited back to have grip tests again after their operation. No aspect of the study will prevent a patient from receiving their normal National Health Service (NHS) care.

DETAILED DESCRIPTION:
RESEARCH QUESTIONS

This study will ask important questions about CTS that builds on previous research in the field. The research questions are:

* How is precision pinch grip force affected by CTS throughout the activity of picking up and replacing an object, for a range of CTS severities, especially in more severe CTS?
* How is precision pinch grip force affected in patients with CTS when picking up objects of different weights?
* How is precision pinch grip force affected in patients with CTS when the frictional properties of the skin-device interface are altered?
* How does precision pinch grip force in CTS alter after a sudden increase in downward load force?
* How do these parameters change after surgical treatment of CTS?

CLINICAL IMPLICATIONS AND STUDY JUSTIFICATION Answers to the above questions will inform understanding of both precision pinch grip force control, and CTS.

Patients with CTS drop things, and the investigators feel that impaired hand function in CTS is related to poor grip control.

Previous authors have recognised that pinch grip force is affected by in CTS (Hsu et al. 2013). The investigators intend to extend this work by showing how other aspects of force control are altered in CTS throughout the action of picking an object up, and how they correlate with CTS severity. This will allow us to use different readings taken during a pinch grip test to assess CTS severity. This will also reveal how heavy objects may have a greater adverse affect on grip control in CTS patients.

If successful, pinch grip testing could form a table-top test for CTS and nerve injury evaluation and may allow better patient selection for surgery.

The investigators will also account for skin hydration, as sweating is impaired in CTS, and rarely accounted for in previous work. (This has since been abandoned mid-study). When examining how friction impacts on precision pinch force in CTS, investigators may inform understanding of how investigators could design occupational aids for those with median nerve problems.

Investigating how patients with CTS compensate when an object they are holding suddenly changes weight, will help us understand reflexes that are co-ordinated by the hand, and may help us in working towards rehabilitating patients after nerve injury affecting the upper limb.

We currently do not have good evidence about which patients should have surgery in CTS or whether surgery restores the hand function that was lost when patients were suffering with CTS. Investigating what happens to the above after surgery, may show us the best time to operate on these patients, which patients we should prioritise and whether surgery actually improves pinch force control post-operatively.

DEVELOPMENT OF RESEARCH PROPOSAL This research proposal has been formulated with experience from senior hand surgeons and multidisciplinary team professionals at a regional hand surgery centre with an active research base (The Birmingham Hand Centre, University Hospitals Birmingham, UK). Consultation has been carried out with the attached University of Birmingham's Department of School of Psychology. A lead collaborator is the department's Professor of Human Movement.

RECRUITMENT Patients with CTS will routinely be referred to the investigators' centre for assessment and treatment of CTS. They would normally be referred to the centre by their GP, receive an appointment letter and attend the hospital. They would then be evaluated clinically and with nerve conduction tests. This may be by a hand surgery consultant or member of the hand team. Patients may then receive a date for surgery and would be followed up if necessary. The Principle Investigator and one Local Collaborator are both consultant hand surgeons who would receive referrals and see these patients in clinic.

Recruitment will occur at one of the following points;

1. At the point at which patients are referred to the Principle Investigator, patients will be offered the chance to participate in their appointment letter which will contain the Participant Information Sheet. This will be further assessed upon presentation to clinic.
2. Some patients are listed for surgery without being seen in the investigators' research clinic, but are suitable for inclusion and are therefore "missed". The investigators intend to recruit these patients already listed for operations for carpal tunnel syndrome on the day of surgery. The Chief Investigator will approach these patients on the day of their operation to seek their permission to carry out pinch-grip testing before surgery. Patients would receive the Patient Information Sheet from the Chief Investigator, and would be consented for study inclusion and tested within the Ambulatory Care Unit of the hospital whilst waiting for their operation. There would be no alteration to their normal care and certainly no delay to their operation.

Recruitment will not affect normal NHS (National Health Service) care in any way. Very limited data (if any) can be collected until the point at which the patient attends for their normal NHS (National Health Service) appointment. If they choose not to take part, they can attend their normal NHS (National Health Service) appointment without the need to undergo grip testing. No therapeutic promises are made by the Participant Information Sheet.

Recruitment of "control" participants; Healthy, age-gender matched controls will be invited from the staff and student body from the University of Birmingham to take part in the pinch grip testing exercise alone to act as a control group.

The investigators will request responses from university members aged 18-80. Potential participants will be invited to take part by email circulated to staff and students. Interested participants who respond by email will receive the full Participant Information Sheet for Controls. This will specify that the only information collected will comprise their age, gender, hand dominance and the grip test data (GP Contact details will be stored anonymously in the case that incidental findings are discovered and warrant action).

They will be invited to attend the University Hospital Birmingham where grip strength tests are performed to undergo testing according to the same protocol outlined for the patient group. This is the point at which consent will be taken by the Chief Investigator or an appropriate member of the research team.

The sample size will be determined by the power analysis run at the beginning of the study, but is expected to comprise 50 patients.

This recruitment process was noted mid-study to be failing to recruit age-matched controls. As an alternative, patients were matched with their own, contralateral hand if it was free of symptoms of CTS.

No formal power analysis took place, as the minimally important clinical difference was not known.

INCLUSION/ EXCLUSION CRITERIA

Inclusion criteria:

Patients with symptomatic, idiopathic CTS (as affirmed by clinical examination and NCS) presenting to clinic Aged between 18 and 80 years In contrast to other studies the investigators would include patients with; Previous upper limb injuries Previous upper limb surgery or CTS intervention (e.g. steroid injections) Diabetes mellitus Any other upper limb nerve neuropathies or upper limb neurology Upper limb musculoskeletal degenerative disease (osteoarthritis) Thyroid disease, (Zhang et al. 2011). This will create a pragmatic study design, generalisable to a wider population in clinical practice.

Exclusion Criteria:

Central neurological or psychiatric disease Visual impairment or any other impairment that would interfere with the patient's ability to perform the study tests Pregnant patients. (Criteria based on prior research (Zhang et al. 2011)).

CONSENT The consent form is that suggested by the Medical Reseach Council (MRC) Health Research Authority and the Participant Information Sheet follows their guidelines. Both will be distributed in appointment letters sent to patients. Informed consent to participate will be confirmed during the original clinic appointment. Members of the hand team consent patients for operations almost daily, and should be fully familiar with assessment of capacity and understanding the ethical principles underpinning informed consent. Consent will be obtained by the Chief Investigator (CI). The study will not include the assessment of children or vulnerable adults

RISKS, BURDENS AND BENEFITS Patients will be informed of all risks and benefits anticipated using the Participant Information Sheet. The investigators cannot guarantee any treatment benefits and do not yet know what the results will show. However, patients will be helping us understand an important problem affecting many other similar patients. These patients may benefit from this research in the future. With their consent, a lay summary will be circulated to the patients and controls after the completion of the study to inform them of the results of the work. They will be consented for this and informed of this in the participation sheets. Their preferred contact details will be stored separately in the index spreadsheet on the trust computer system and will not be linked with clinical data.

The intent is to carry out pinch grip force testing on CTS patients. This will add to the time patients are asked to stay in clinic by about 30 minutes. They will be fully informed and asked whether they wish to participate, prior to being invited to take part in precision pinch grip testing. This will not affect their access to assessment or treatment of their CTS.

The intent is to test precision pinch grip testing with a custom built device being developed by the University of Birmingham. This device is based on those already used by Zhang and Hsu et al, and is not anticipated to pose any risk of harm to the patient. The investigators do not know of any side effects that there may be from the grip test. Patients may find their hand to be a little tired after the test; however this should not last long and should not be severe. The investigators think the risk of injury posed to patients by the grip device is very small. The investigating team will have trialed the device on healthy volunteering members of the research team prior to use in the study.

The investigators do not think that there will be any risks; including but not limited to psychological or physical harm, posed by the study that fall outside the risks inherent in normal clinical care.

Confidentiality breech is extremely unlikely, as all information will be stored on NHS (National Health Service) trust computers, however the investigators acknowledge this risk. Only clinicians involved in patient care or researchers from within the study team will have access to patients' clinical details. Patients will be consented to allow non-clinical members of the research team (university staff) access to essential information for the study; however this information will be kept to an absolute minimum. For example, if a researcher performs the "pinch-grip" test, it is fair to assume that researcher will become aware that the patient has a diagnosis of CTS. Patients will have been consented for this.

The burden of patients being requested to attend three subsequent follow-up appointments is acknowledged, however the above benefits patients may feel in contributing to this study will encourage them to attend.

The study sponsor (UHB) will be updated throughout, with special emphasis placed on drawing attention to any risks or burdens that emerge after the start of the study.

The above risks are all conveyed in the Participant Information Sheet.

CONFIDENTIALITY Confidentiality Principles Principle 1: The purposes of obtaining patient information are outlined above. Principle 2 and 3: Person-identifiable data will not be collected. Participants will be identified by UHB Patient Number.

Principle 4: Access to person-identifiable data will be limited to members of the treating clinical team only. If non-clinical collaborators perform the precision pinch-grip test in clinic, they will not have access to patient-identifiable clinical details, during the test or afterwards during analysis.

Principle 5 and 6: All clinical team members are aware of their commitment to confidentiality and the law.

The investigators do not anticipate that these principles will need to be breached in order to prevent serious patient harm. If however, this situation arises, it will be discussed between the Chief and Principle Investigators, the relevant authorities will be contacted for advice and action taken whilst taking all steps to safely inform affected patients as early as possible.

CONFLICTS OF INTEREST The Principle or Chief Investigators will be involved in clinical evaluation of CTS patients at their appointment. Special care will be taken to ensure patients are aware that study participation does not affect their normal care in any way. Care will be taken to avoid any form of coercion. The Principle or Chief Investigators may also perform surgical treatment on appropriate patients, however this is separate to the study and should not affect care in any way. Effort will be made to ensure patients are not coerced into returning for follow-up grip testing after their operation. Patients may wish to attend extra follow-up appointments. At the end of the study, patients are discharged back to the care of their GP, to be referred back if any concerns arise (as is normal practice). Participants will be aware that they will not know the results of their grip tests, but the intent will be to publish a full paper within twelve months.

HUMAN TISSUE Non- applicable

OTHER ETHICAL ISSUES The intent is to carry out pinch grip force testing on CTS patients. This will add to the time patients are asked to stay in clinic. They will be fully informed and asked whether they wish to participate, prior to being invited to take part in precision pinch grip testing. This will not affect their access to assessment or treatment of their CTS.

The intent is to test precision pinch grip testing with a custom built device being developed by the University of Birmingham. This device is based on those already used by Zhang and Hsu et al, and is not anticipated to pose any risk of harm to the patient.

OTHER LEGAL ISSUES As the device is being custom-built by the University of Birmingham, intellectual property rights are being addressed by the department developing the device, with a view to drawing up a confidentiality agreement, although this is not a pre-requisite to commencing the trial.

OTHER MANAGEMENT ISSUES This intention is to set-up an National Health Service (NHS) clinic of back-to-back CTS patients, who will have a clinical assessment, followed by nerve conduction studies, followed by pinch grip assessment. This will require logistic planning, however this will be co-ordinated internally through UHB and will make the process clear to patients when they are recruited to the study via the Participant Information Sheet.

ELIGIBILITY:
Inclusion criteria:

Patients with symptomatic, idiopathic CTS (as affirmed by clinical examination and NCS) presenting to clinic Aged between 18 and 80 years In contrast to other studies the investigators would include patients with; Previous upper limb injuries Previous upper limb surgery or CTS intervention (e.g. steroid injections) Diabetes mellitus Any other upper limb nerve neuropathies or upper limb neurology Upper limb musculoskeletal degenerative disease (osteoarthritis) Thyroid disease, (Zhang et al. 2011). This will create a pragmatic study design, generalisable to a wider population in clinical practice.

Exclusion Criteria:

Central neurological or psychiatric disease Visual impairment or any other impairment that would interfere with the patient's ability to perform the study tests Pregnant patients. (Criteria based on prior research (Zhang et al. 2011)).

Control population is as previously specified.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: See inclusion/ exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Change in Precision Pinch Grip Force measured during a pinch-hold up activity over time during follow-up | Assessed at initial outpatient appointment, at 3, 6 and 12 months
  Precision pinch grip force will be measured over time during a pinch-hold up activity. Change in this force will be observed over time at 3, 6 and 12 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Power, FRCS, Principal Investigator — University Hospital Birmingham
Locations (1):
- University Hospitals Birmingham Queen Elizabeth, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Background] Zhang W, Johnston JA, Ross MA, Smith AA, Coakley BJ, Gleason EA, Dueck AC, Santello M. Effects of carpal tunnel syndrome on adaptation of multi-digit forces to object weight for whole-hand manipulation. PLoS One. 2011;6(11):e27715. doi: 10.1371/journal.pone.0027715. Epub 2011 Nov 16. PMID 22110738
- [Background] Zhang W, Johnston JA, Ross MA, Sanniec K, Gleason EA, Dueck AC, Santello M. Effects of carpal tunnel syndrome on dexterous manipulation are grip type-dependent. PLoS One. 2013;8(1):e53751. doi: 10.1371/journal.pone.0053751. Epub 2013 Jan 10. PMID 23326498
- [Background] Padua L, Lo Monaco M, Padua R, Gregori B, Tonali P. Neurophysiological classification of carpal tunnel syndrome: assessment of 600 symptomatic hands. Ital J Neurol Sci. 1997 Jun;18(3):145-50. doi: 10.1007/BF02048482. PMID 9241561
- [Background] Yen WJ, Kuo YL, Kuo LC, Chen SM, Kuan TS, Hsu HY. Precision pinch performance in patients with sensory deficits of the median nerve at the carpal tunnel. Motor Control. 2014 Jan;18(1):29-43. doi: 10.1123/mc.2013-0004. PMID 24496877
- [Background] Verghese J, Galanopoulou AS, Herskovitz S. Autonomic dysfunction in idiopathic carpal tunnel syndrome. Muscle Nerve. 2000 Aug;23(8):1209-13. doi: 10.1002/1097-4598(200008)23:83.0.co;2-#. PMID 10918257